CLINICAL TRIAL: NCT01509417
Title: Prospective Randomized Trial Evaluating the Feeding Regimen After Pyloromyotomy.
Brief Title: Different Feeding Methods After Pyloromyotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10 05-101
Record Dates: First submitted 2011-12-14; First posted 2012-01-13 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Emesis
Keywords: pyloric stenosis
MeSH Terms: conditions — Vomiting; Pyloric Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ad lib feeding (Experimental): ad lib feedings following pyloromyotomy
  Interventions: Other: ad lib feedings after pyloromyotomy; Other: FLAP diet after pyloromyotomy
- FLAP diet after pyloromyotomy (Active Comparator): FLAP diet after pyloromyotomy
  Interventions: Other: FLAP diet after pyloromyotomy

INTERVENTIONS:
Other: ad lib feedings after pyloromyotomy — ad lib feedings after pyloromyotomy
  Other Names: post surgical refeeding ad lib
  Arms: Ad lib feeding
Other: FLAP diet after pyloromyotomy — FLAP diet after pyloromyotomy
  Other Names: Post surgical FLAP refeeding

SUMMARY:
The objective of this study is to scientifically evaluate the ability to discharge patients based on feeding schedule comparing ad lib feeds to our current scheduled regimen.

The hypothesis is that patients may be able to be discharged sooner with ad lib feeds.

DETAILED DESCRIPTION:
Hypertrophic pyloric stenosis is a common disease occurring in 2 per 1,000 live births1. Pyloric stenosis is a hypertrophy of the pyloric muscle which prevents emptying of the stomach leading to gastric outlet obstruction. The vomiting that ensues becomes projectile and results in severe dehydration. Traditionally this has been repaired with the pyloromyotomy via a transverse incision in the right upper quadrant. In the last decade the investigators have started doing the same procedure laparoscopically. Most institutions follow similar guidelines as to what constitutes a hypertrophic pyloric channel, initial electrolyte management and resuscitation prior to surgery, as well as the pyloromyotomy (either open or laparoscopically).

Historically patients were fed the day after surgery, then 6 hours, and currently the investigators wait 2 hours after surgery to start feeds. The investigators go through a protocol of 2 rounds of clear liquids, 2 rounds of half strength formula/breast milk then 2 rounds of full strength. Some centers have advocated ad lib feeds where babies go straight to full strength as tolerated when awake from the operation.

Institutional variability is even further confounded by individual attending variability in some instances. Recent articles in the past two decades still prove that no consensus has been found. Some institutions profess that Ad Libitum feeding is both cost-effective as well as safe, but very few institutions to our knowledge follow this mantra. Others demand that no feeds should be started within 4 hours post surgery stating that the increased vomiting associated with this early feeding regimen actually prolongs the time to full feeds due to anxiety and discomfort. What has been shown is that no matter whether patients start 4 hours post surgery or wait 18 hours the time to full feeds is the same. All of these studies are hindered by the fact that they all have retrospective components to their design.

What has also been propagated in two recent retrospective reviews is the implementation of clinical pathways as well as standardized feeding regimens. Both of these showed a decrease in length of stay postoperatively as well as hospital costs.

At our institution a clinical pathway and feeding regimen has been implemented. The feeding regimen contrary to some of the previously quoted papers starts at 2 hours with sequential feeding increases. A prospectively acquired dataset at our institution has shown that emesis is correlated to the degree of dehydration of the child prior to surgery even with all the children being on the same clinical pathway.

What all of these studies show us is that as a profession, Pediatric Surgery does not have the proper evidence to support any one post-op feeding regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with pyloric stenosis and scheduled for laparoscopic pyloromyotomy. -

Exclusion Criteria:

* Open procedures
* Patient has alternative diagnosis that would affect feeding (like mucosal perforation)

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | up to 10 days

SECONDARY OUTCOMES:
number of emeses during stay | up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital and Clinics
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States